CLINICAL TRIAL: NCT06380127
Title: Feasibility and Effectiveness of a 12-week Concurrent Exercise Training on Physical Performance, Muscular Strength and Circulating Myokines in Frail Older Adults Living in Nursing Homes: a Cluster Randomized Crossover Trial
Brief Title: Feasibility and Effectiveness of Concurrent Exercise Training on Frail Older Adults Living in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Maria Joana Carvalho, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CEFADE012021
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Frailty
Keywords: Frail; Exercise; Concurrent training; Long-term care; Myokines
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The trial will follow a 28-week crossover design: 12 weeks for the first intervention period, a 4-week washout, and another 12 weeks for the second intervention period. Nursing homes (clusters) were randomized into sequences (AB or BA), where intervention A involve concurrent exercise training, and B is usual care.
  Data collection will occurre at four points: baseline, post-first intervention period, post-washout/pre-second intervention period and post-crossover.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Progressive concurrent exercise training
  Interventions: Behavioral: Exercise training
- Usual Care (No Intervention): The usual care

INTERVENTIONS:
Behavioral: Exercise training — The exercise intervention will take place at the nursing homes and consists of 12 weeks of supervised concurrent exercise training, performed thrice weekly on nonconsecutive days to avoid overtraining and fatigue. Each session will last 50-60 min and consist of a warm-up, resistance plus aerobic training, and a 5-min cool-down period. The resistance training will comprise 2-3 sets of 10 to 15 repetitions with a load equivalent to 40 to 70% of the 1-repetition maximum (1RM) for upper (i.e., bicep curl) and lower body exercises (i.e., seated knee extension). The sit-to-stand exercise will be performed as fast as possible according to each participant's capacity without external load. The recovery between sets is between 1 and 2 min. Afterwards, participants will perform walking exercises with changes in pace and direction. The duration of the aerobic training will progress from 5-10 min duration in the first weeks to 10-15 min. The sessions will end with stretching exercises.The exercise
  Arms: Exercise

SUMMARY:
The present study is a crossover randomized controlled trial that aims to investigate the effects of concurrent exercise training over usual care on physical performance, muscle strength, and myokines concentrations in frail older adults living in nursing homes.The main questions it aims to answer is: Can a 12-week exercise intervention provide beneficial effects on physical performance, muscle strength and myokines among the most frail participants? Researchers will compare this intervention to usual care. Nursing homes (comprising participants) will be randomly assigned to a sequence of interventions (AB or BA), being A -exercise and B usual care. Participants will be assessed before and after each intervention.

DETAILED DESCRIPTION:
The present study is a crossover randomized controlled trial that aims to investigate the effectiveness of a concurrent exercise training over usual care on physical performance, muscle strength, and myokines concentrations in frail older adults living in nursing homes. Nursing homes will be randomly assigned to receive a sequence of interventions (AB or BA), being A -exercise and B usual care. Participants will receive a 12-weeks of either exercise intervention or usual care. A 4-week washout period will be conducted between interventions. Participants will assessed before and after each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Classified as frail according to the Fried criteria (e.g., frailty phenotype ≥ 3 criteria);
* Not having participated in any exercise intervention for the last 3 months;
* Being able to ambulate (with/without assistance).

Exclusion Criteria:

* Any contraindication that could affect physical exercise performance or testing procedures, including terminal illness, uncontrolled disease or other unstable medical condition;
* Bone fracture in the past three months;
* having a short physical performance battery score (SPPB) < 3.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Short Physical Performance Battery (SPBB) | Assessment at baseline and immediately after 12 weeks of intervention, in each period.
  The Short Physical Performance Battery (SPPB) is a standardised assessment tool of lower limb function, testing 3 dimensions: standing balance, walking speed, and chair stands. Each component is scored between 0-4, total score from 0 (poor performance) to 12 (best performance).

SECONDARY OUTCOMES:
Change from Baseline on Handgrip test | Assessment at baseline and immediately after 12 weeks of intervention, in each period
  Handgrip strength will be obtained with a Jamar Plus + Digital hand dynamometer (Sammons Preston Inc., Bolingbrook, Illinois, USA).Measurements will be carried out following the American Society of Hand Therapists recommendations, and each participant will perform three attempts with a pause of 15s between trials
Change from baseline on isokinetic knee strength | Change from baseline and 12 weeks in each intervention, in both periods
  The dynamic concentric muscle strength of the knee flexors and extensors will be measured on an isokinetic dynamometer (Biodex System 4 Pro; Biodex, Shirley, NY).The measurements will follow the manufacturer's instructions for knee extension/flexion at the angular velocity of 60/s (1.05 rad/s). After a few repetitions for familiarization, each participant will perform three maximal repetitions at 60/s with their preferred leg.
Change from Baseline on circulating levels of myostatin | Change from baseline and 12 weeks in each intervention, in both periods
  Determination of myostatin levels in serum.
Change from Baseline on circulating levels of Decorin | Assessment at baseline and immediately after 12 weeks of intervention, in each period
  Determination of decorin levels in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Carvalho, PhD, Principal Investigator — CIAFEL
Locations (1):
- Faculty of Sports, University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barros D, Silva-Fernandes A, Martins S, Guerreiro S, Magalhaes J, Carvalho J, Marques EA. Feasibility and Effectiveness of a 12-Week Concurrent Exercise Training on Physical Performance, Muscular Strength, and Myokines in Frail Individuals Living in Nursing Homes: A Cluster Randomized Crossover Trial. J Am Med Dir Assoc. 2024 Nov;25(11):105271. doi: 10.1016/j.jamda.2024.105271. Epub 2024 Sep 19. PMID 39305935